CLINICAL TRIAL: NCT02748720
Title: Impact of Measurement of Respiratory Dynamics During Birth Stabilization in Preterm Infants Less Than 32+6/7 Weeks Gestation
Brief Title: Respiratory Dynamics During Birth Stabilization in Preterm Infants Less Than 32+6/7 Weeks Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Sanchez Luna (Other)
Responsible Party: Sponsor-Investigator, Manuel Sanchez Luna, Dr, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-05
Record Dates: First submitted 2016-04-04; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Infant, Premature
Keywords: Premature; Respiratory Function Monitor
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFM Visible (Experimental): Patients will be randomize in other Group 1, where these parameters (from the device Respiratory Function Monitor) of lung mechanics would be visible by the rescuer (the usual parameters of PIP and PEEP will be visible). We adapt or change PIP using visible TVe.
  Interventions: Other: RFM (device) Visible
- RFM No Visible (No Intervention): Patients will be randomize in a Group 2, where the parameters of TVe and respiratory flow would not be visible by the rescuer (the usual parameters of PIP and PEEP will be visible). Always, in both groups, current recommendations ventilation measures included in cardiopulmonary resuscitation of newborns of the Spanish Society of Neonatology, based on international recommendations (1-3.5) apply. In turn, the results analyzed in two subgroups between 24 and 27 + 6 weeks gestational age and 28 to 32 + 6 weeks

INTERVENTIONS:
Other: RFM (device) Visible — Will measure the expire tidal volume, end tidal CO2 and peak pressure changes according to clinical improvement and tidal volume
  Arms: RFM Visible

SUMMARY:
Approximately 50% of preterm infants less than 32 weeks require respiratory assistance at the time of transition at birth. For that stabilization during resuscitation is successful, it is essential for proper ventilation. This transition is performed with non-invasive respiratory support and administration of positive pressure ventilation to establish adequate functional residual capacity. The problem is that a peak inspiratory fixed during ventilation, and adequate tidal volume is assumed, but usually not measured, unable to correct the peak pressure to optimize ventilation and reduce lung damage. In addition, frequent adverse events may hinder or impair the effectiveness of the ventilation, with the consequent deterioration in the prognosis of the newborn.

DETAILED DESCRIPTION:
HYPOTHESIS The ability to visualize the parameters and curves respiratory flow, tidal volume and air pressure by respiratory monitoring with MFR during cardiopulmonary resuscitation in newborns in the delivery room, decreases at least 10% surfactant need in first 72 hours of life.

EVALUATION Data collection will be made prospectively. Investigators will measure the parameters of lung mechanics (tidal volume expiratory airflow (TVe), peak inspiratory pressure (PIP), pressure at the end of exhalation (PEEP), inspiratory time (iT)), in each of inflations administered to preterm with VPP or during the administration of continuous positive airway pressure (CPAP) in spontaneous breathing, in the first 10 minutes after birth, recording the air leakage through the mask and obstructions. Investigators also measure parameters of respiratory status and hemodynamic (FIO 2, oxygen saturation, end tidal CO2, respiratory rate, heart rate), patient monitoring during the implementation of the protocol, blood gases, manipulations of the airway during intervention and the onset of complications.

Patients will be randomize in a Group 1, where these parameters of lung mechanics would be visible and other Group 2, where the parameters of TVe and respiratory flow would not be visible by the rescuer (the usual parameters of PIP and PEEP will be visible). Always, in both groups, current recommendations ventilation measures included in cardiopulmonary resuscitation of newborns of the Spanish Society of Neonatology, based on international recommendations (1-3.5) apply. In turn, the results analyzed in two subgroups between 24 and 27 + 6 weeks gestational age and 28 to 32 + 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* infants less than 32+6/7 weeks gestational age, birth requiring stabilization with VPP or CPAP in the delivery room.

Exclusion Criteria:

* Congenital Malformations or Chromosomal Aberrations
* Less Than 22 Weeks
* Birth-weight less Than the Third Percentile for Gestational Age According to Spanish Curve
* Severe Perinatal Asphyxia (Apgar Score of 0-3 More Than 5 Min, Cord Blood ph<7.00)
* reanimation unrecorded with video
* no obtained informed consent

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduce the need for surfactant. | through study completion, an average of 3 days
  The aim of this study is to investigate whether the use of MFR during resuscitation of preterm (24-32 + 6 weeks) reduce the need for surfactant.

SECONDARY OUTCOMES:
Need for intubation and intermittent mechanical ventilation (iMV) | through study completion, an average of 3 days
  Avoid intubation and Invasive Mechanical Ventilation in the next three days.
Incidence of dysplasia bronchopulmonary | through study completion, an average of 1 year
  Reduce incidence of dysplasia bronchopulmonary
CPAP on admission to NICU | through study completion, an average of 1 day
  Number of newborn with CPAP on admission to NICU
Incidence of mortality | through study completion, an average of 1 year
Measure and get desired tidal volume to optimize resuscitation | through study completion, an average of 1 year
Number of leaks and obstruction during ventilation mask | through study completion, an average of 1 day
  The aim of this study is to investigate whether the use of MFR during resuscitation of preterm (24-32 + 6 weeks) reduce number of leaks and obstruction during mask ventilation and improves and set the desired tidal volume to optimize resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Zeballos, MD, Principal Investigator — Gregorio Marañón Hospital
Locations (1):
- HGU Gregorio Marañón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No